CLINICAL TRIAL: NCT00410319
Title: Information or Physical Activity for Chronic LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VF 20040016
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Behavioral: Fear-reducing Information
Behavioral: Symptom-based exercise

SUMMARY:
The purpose of this study is to compare a specific fear-reducing information with symptom-based exercise

ELIGIBILITY:
Inclusion Criteria:

* Daily LBP, dominating over possible pain in leg or other joints/muscles
* Pain og > 4 (scale 0-10) for more than 4 months

Exclusion Criteria:

* Cancer, inflammatory disease, previous back surgery, pregnancy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bendix, dr.med prof, Study Director — University of Southern Denmark

REFERENCES:
- [Derived] Sorensen PH, Bendix T, Manniche C, Korsholm L, Lemvigh D, Indahl A. An educational approach based on a non-injury model compared with individual symptom-based physical training in chronic LBP. A pragmatic, randomised trial with a one-year follow-up. BMC Musculoskelet Disord. 2010 Sep 17;11:212. doi: 10.1186/1471-2474-11-212. PMID 20849601